CLINICAL TRIAL: NCT06063148
Title: Neonatal Pulse Oximetry Disparities Due to Skin Pigmentation
Acronym: Neo-PODS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1840688
Record Dates: First submitted 2023-08-02; First posted 2023-10-02 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Skin Pigment; Pulse Oximetry
MeSH Terms: conditions — Pigmentation Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Enrolled Participant (Experimental): During routine arterial blood gas sampling, a coordinator will measure SpO2 from a similar extremity. SpO2 data will be recorded using Masimo Radical-7 oximeters. To minimize ambient light interference or optical cross talk from other SpO2 sensors, all the SpO2 sensors will be fully shielded with cloth wraps provided by Masimo. Each enrolled infant will undergo simultaneous blood gas sampling and SpO2 measurement for each routine blood gas collected. Up to a total of 10 SpO2 measurements will be collected, paired with 10 blood gas samples collected as part of routine care, though We anticipate about 3 paired samples (SaO2 and SpO2) per enrolled infant.
  Interventions: Device: Enrolled Participant

INTERVENTIONS:
Device: Enrolled Participant — Participant will undergo at most 10 SpO2 measurements paired with at most 10 routine blood gas samples.

SUMMARY:
The goal of this clinical trial is to determine if pulse oximeters show an SaO2-SpO2 discrepancy that correlates with skin pigmentation such that pulse oximetry will overestimate oxygenation in newborns with darker skin. The main questions it aims to answer is if SaO2-SpO2 discrepancy varies with the degree of skin pigmentation among neonates, if gestational age has an influence on SaO2-SpO2 discrepancy, and if packed red blood cell (PRBC) transfusion has an influence on SaO2-SpO2 discrepancy in newborns with various degrees of light and dark skin. Researchers will compare SaO2 and SpO2 values in neonates of various skin pigmentation.

DETAILED DESCRIPTION:
Investigators will use a multicenter prospective cohort approach to measure SpO2 and SaO2 simultaneously in newborns of varying degrees of light and dark skin. The investigators will enroll 163 newborns of varying degrees of light and dark skin to assess the impact of skin pigmentation on the accuracy of pulse oximetry. Data collection will occur during routine blood samples and will involve simultaneous measurement of oxygen saturation by pulse oximetry and additional data extraction from the EHR. The study consists of 4 main components: (1) Skin pigment classification (2) Race and ethnicity classification (3) SpO2 measurement collection (4) EMR data collection (including newborn screen hemoglobin type assessment and transfusion records). After adjusting for SaO2, the SaO2-SpO2 discrepancy will correlate with skin pigmentation such that pulse oximetry will overestimate oxygenation in newborns with darker skin. The distribution of SaO2-SpO2 discrepancy will have more variance in the newborns with darker skin.

ELIGIBILITY:
Inclusion Criteria:

* Newborns postnatal age < 10 days admitted to intensive care unit
* Presence of arterial catheter or undergoing arterial stick blood gas sampling

Exclusion Criteria:

* <26 weeks corrected gestational age (After May 2024, infants <26 weeks corrected GA were excluded due to skin irritation with sensor removal, those enrolled earlier were included in the analysis)
* Presence of abnormal hemoglobin (including methemoglobin > 3%) - likely to only be known after enrolled and the blood gas is obtained
* Those in whom SpO2 cannot be measured in the same extremity as the arterial catheter.

Max Age: 10 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 163 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Determine if SaO2-SpO2 discrepancy varies with the degree of skin pigmentation among neonates. | Through study completion, about 2 years
  Using a prospective cohort of 163 newborns, the investigators will calculate simultaneous SaO2-SpO2 discrepancy and correlate it with a measure of skin pigmentation (melanin index: Fitzpatrick Scale, Massey-Martin scale and ITA: individual Typology Angle) among neonates with and without hypoxemia.
Determine the influence of packed red blood cell (PRBC) transfusion on SaO2-SpO2 discrepancy in newborns with various degrees of light and dark skin. | Through study completion, about 2 years
  Many infants in the NICU setting are transfused PRBC with hemoglobin A, which shifts the oxygen-hemoglobin dissociation curve to the right. While the effect of this shift on pulse oximetry is studied, the combined impact of skin pigmentation and transfusion is not known. The investigators will test the hypothesis that PRBC transfusion increases the impact of skin pigmentation on SaO2- SpO2 discrepancy. The investigators will calculate the SaO2-SpO2 discrepancy and correlate it with the skin pigmentation measurement and frequency of PRBC transfusion.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - UC Davis Health, Sacramento, California
  - University of Mississippi Medical Center, Jackson, Mississippi

IPD SHARING:
Plan to Share IPD: No